CLINICAL TRIAL: NCT03475121
Title: GALOP II Protocol for the Treatment of Unilateral Retinoblastoma
Brief Title: Treatment Protocol for Non-Metastatic Unilateral Retinoblastoma
Acronym: RbGALOP2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital JP Garrahan (Other Government)
Responsible Party: Principal Investigator, Pedro Zubizarreta, MD, Head Hematology and Oncology Department, Hospital JP Garrahan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1031. Retinoblastoma GALOP 2
Record Dates: First submitted 2018-03-12; First posted 2018-03-23 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Unilateral Retinoblastoma
MeSH Terms: interventions — Drug Therapy, Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low Risk Patients (Experimental): Patients with IRSS stage I, pT1, pT2 and pT3 stage will not receive adjuvant therapy
  Interventions: Other: No Adjuvant Therapy
- Higher Risk Patients (Experimental): Patients with IRSS stage I, pT3b, pT3c, pT3d will receive 6 cycles of adjuvant chemotherapy plus 6 doses of intrathecal topotecan
  Interventions: Combination Product: Combination Chemotherapy plus Intrathecal Topotecan
- Stage II Patients (Experimental): Patients with Stage II (pT4) will receive 6 cycles of adjuvant chemotherapy plus 6 doses of intrathecal topotecan and orbital radiotherapy
  Interventions: Combination Product: Higher Dose Combination Chemotherapy plus Intrathecal Topotecan and Orbital Radiotherapy
- Patients with buphthalmus (Experimental): Patients with buphthalmus (cT3c, cT3e) will receive 2 cycles of neo-adjuvant chemotherapy plus 6 doses of intrathecal topotecan followed by secondary enucleation and 6 cycles of adjuvant chemotherapy.
  Interventions: Combination Product: Higher Dose Combination Chemotherapy plus Intrathecal Topotecan

INTERVENTIONS:
Combination Product: Combination Chemotherapy plus Intrathecal Topotecan — Adjuvant chemotherapy with a reduced dose (compared to GALOP I protocol) of carboplatin
  Arms: Higher Risk Patients
Combination Product: Higher Dose Combination Chemotherapy plus Intrathecal Topotecan — GALOP I-based systemic adjuvant therapy plus intrathecal topotecan
  Arms: Patients with buphthalmus
Combination Product: Higher Dose Combination Chemotherapy plus Intrathecal Topotecan and Orbital Radiotherapy — GALOP I-based systemic adjuvant therapy plus intrathecal topotecan and orbital radiotherapy (45 Gy) up to chiasm
  Arms: Stage II Patients
Other: No Adjuvant Therapy — Patients will not receive any adjuvant therapy after enucleation of the affected eye.
  Arms: Low Risk Patients

SUMMARY:
This protocol provides guidelines for the management of non-metastatic unilateral retinoblastoma and introduces an innovative adjuvant therapy for higher risk patients based upon the results of the Grupo de America Latina de Oncologia Pediatrica (GALOP) I study. Conservative therapy will be not protocolized.

DETAILED DESCRIPTION:
Patients with non-metastatic retinoblastoma undergoing enucleation will be staged using the American Joint Committee on Cancer (AJCC), version 8, Tumor, Node, Metastasis (TNM)- H system and the International Retinoblastoma Staging System (IRSS). IRSS stage I patients recognized as higher risk will be assigned for adjuvant therapy. Those with standard risk will not receive adjuvant therapy after enucleation. Higher risk patients are defined as those with pathological retrolaminar optic nerve invasion and-or any degree of scleral invasion (pT3b, pT3c, pT3d). Based on the results of the GALOP I protocol, they will receive a reduced dose adjuvant chemotherapy regimen with 3 cycles of alternating cyclophosphamide, vincristine and idarubicin alternating with another 3 cycles of carboplatin and etoposide. Six doses of intrathecal topotecan will be given. Patients presenting with severe buphthalmia (cT3c-cT3e) will receive neo-adjuvant therapy with the same intensive regimen but including a higher dose of carboplatin as per GALOP I protocol plus intrathecal topotecan and secondary enucleation followed by adjuvant chemotherapy for a total of 8 cycles. Stage II patients (pT4) will receive the same adjuvant regimen plus orbital radiotherapy (45 cGy).

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of retinoblastoma confirmed at participating institutions
* Ophthalmological diagnosis of unilateral retinoblastoma in patients undergoing conservative therapy.
* No prior therapy for retinoblastoma
* Lansky Performance Scale greater or equal to 50
* Normal organ function in those patients assigned for chemotherapy
* Signed informed consent

Exclusion Criteria:

* Patients with unilateral retinoblastoma and germline mutations of the Rb1 gene or family history for retinoblastoma

Ages: 0 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Rate of extraocular relapses | 3 years
  Number of participants experiencing extraocular relapse
Evaluation of number of patients experiencing acute, chronic and fatal toxicities | 5 years
  Number of participants experiencing treatment-related adverse effects and mortality as measured by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital JP Garrahan, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No